CLINICAL TRIAL: NCT07362576
Title: Improving the Perinatal Mental Health of Veterans With Serious Mental Illness Through Peer Support
Brief Title: Perinatal Peer Support for Veterans With Serious Mental Illness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSR5-008-24W; CDX 25-003 (Other Grant/Funding Number: VA HSR); IK2RD000606-01A1 (NIH)
Record Dates: First submitted 2025-12-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Persons With Psychiatric Disorders
Keywords: Pregnant Women; Peer Support; Postpartum Care; Veterans Health

STUDY DESIGN:
Intervention Model Description: A feasibility pilot with Veterans with serious mental illness (n=24) enrolled during pregnancy and engaged through approximately 3 months postpartum, randomized to the perinatal peer support intervention or usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus perinatal peer support (Experimental): Participants in this arm will receive the perinatal peer support intervention, delivered by a trained Veteran perinatal peer specialist. They will continue to have access to routinely offered mental health and health services, including but not limited to Maternity Care Coordination, psychiatry, psychotherapy, and/or social work.
  Interventions: Behavioral: Perinatal peer support
- Usual care (No Intervention): Usual care will include access to routinely offered mental health and health services, including but not limited to Maternity Care Coordination, psychiatry, psychotherapy, and/or social work.

INTERVENTIONS:
Behavioral: Perinatal peer support — The final intervention model, components, and timeline will be determined in an iterative process incorporating scientific evidence with input from Veterans, staff, and leadership in Aims 1 and 2. Preliminarily, the intervention is anticipated to begin with perinatal peer specialist contact by week 32 of pregnancy and continue for a duration of ~6 months. Session content may include psychoeducation and assessment of functional goals (e.g., related to employment, relationships, or illness management) and unmet social needs (e.g., housing, childcare, financial). Given that the initial postpartum period is a time of increased need for social support and vulnerability to mental health decline, peer support contact will continue until approximately 3 months postpartum.
  Arms: Usual care plus perinatal peer support

SUMMARY:
Veterans with serious mental illness (SMI) are at high risk of exacerbation of mental illness in pregnancy and postpartum, with consequences including poor pregnancy outcomes, decreased functioning, and impaired child development. Peer support could play a key role in supporting pregnant and postpartum Veterans with SMI. In this study, investigators will develop (Aims 1 and 2) and pilot (Aim 3) a peer specialist-delivered perinatal mental health intervention for Veterans with SMI, drawing from evidence-based models and input from Veterans, key VA clinical staff, and subject matter experts. The intervention will be piloted to assess its feasibility and acceptability, as well as exploratory clinical outcomes including postpartum functioning and mental health symptoms.

DETAILED DESCRIPTION:
There are currently no perinatal mental health interventions designed for or tested among Veterans with SMI. Reach Out, Stay Strong Essentials (ROSE)-a five-session evidence-based psychosocial intervention for prevention of postpartum depression in women without mental illness-is currently being implemented in the VA health care system. To date, ROSE implementers have noted the benefits of the intervention for pregnant Veterans, but have also shared its shortcomings for those with SMI, including its limited attention to current psychiatric symptoms, limited postpartum support, and minimal content related to unmet social or clinical needs.

Peer support-offered by individuals with lived experience of mental illness-is emerging as a key component of VA mental health care, and recent Congressional mandates call for expansion of VA peer support services for women. Perinatal peer support has been shown to improve mental health outcomes in non-SMI populations, but there have been no studies of its effects in women with SMI or Veterans. To address these gaps, the investigators will develop and pilot an adapted, peer specialist-delivered perinatal mental health intervention for Veterans with SMI, blending ROSE with components from evidence-based perinatal and SMI peer support models, and tailored to perinatal Veterans' unique needs and the VA context.

Guided by the Transcreation Framework, an implementation science framework for community-partnered development of behavioral interventions for vulnerable populations, the Specific Aims are to:

Aim 1. Engage Veterans and key VA clinical staff in identifying potential components of a tailored peer support intervention for perinatal Veterans with SMI. Individual semi-structured interviews with pregnant and postpartum Veterans with SMI and VA women's mental health providers will assess the experiences, needs, and care preferences of perinatal Veterans with SMI, as well as desirable intervention components of existing perinatal and peer support interventions. Focus groups with VA Maternity Care Coordinators and women VA peer specialists will also explore intervention components and implementation considerations.

Aim 2. Develop and refine the intervention. Using Delphi methodology, the investigators will present potential intervention components-drawn from ROSE and existing peer support interventions, and accompanied by relevant data from the literature and Aim 1 findings-to an expert panel of VA multilevel constituents to identify final components as well as adaptations to optimize fit to the target population and VA women's health settings. The investigators will then develop the intervention prototype and materials in an iterative process in collaboration with operations partners, women Veteran peer specialists, and mentors.

Aim 3. Assess the feasibility, acceptability, and exploratory outcomes of the intervention in a pilot study. This single-site feasibility pilot will include approximately 24 Veterans with SMI enrolled during pregnancy and engaged through approximately 3 months postpartum, randomized to perinatal peer support or usual care. Mixed methods evaluation will focus on feasibility and acceptability, as well as exploratory clinical (e.g., depression) and service utilization outcomes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant Veterans with serious mental illness

  * a diagnosis of major depressive disorder
  * PTSD
  * bipolar disorder
  * schizophrenia
  * other psychotic disorder

Exclusion Criteria:

* Participants will be enrolled in the outpatient setting, and therefore will not be eligible to enroll while admitted to an inpatient psychiatric unit

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2028-07-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | up to 9 months
  Feasibility of recruitment procedures will be assessed by the percent of eligible Veterans who enroll, and cited reasons for declined participation. Feasibility of retention will be assessed by percent of enrolled participants completing the post-intervention assessment, and cited reasons for study termination or non-completion.
8-item Client Satisfaction Questionnaire (CSQ-8) | within 2 months of intervention completion
  The CSQ-8 will be used to assess acceptability of the intervention to participants. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Participant and provider perspectives | within 2 months of intervention completion
  Qualitative assessment of intervention acceptability, feasibility, and appropriateness will be accomplished through semi-structured post-intervention interviews with participants, peer specialists, and adjacent staff (women's mental health providers, maternity care coordinators).

SECONDARY OUTCOMES:
Barkin Index of Maternal Functioning (BIMF) | up to 9 months
  Postpartum functional status will be assessed using the 20-item BIMF.
24-item Behavior and Symptom Identification Scale (BASIS-24) | up to 9 months
  The BASIS-24 is a widely used, validated instrument capturing degree of distress or impairment, overall and on six subscales (Depression/Functioning, Relationships, Self-Harm, Emotional Lability, Psychosis, and Substance Abuse).
Edinburgh Postnatal Depression Scale (EPDS) | up to 9 months
  The EDPS is a 10-item depression screening tool, validated for use in both pregnancy and postpartum.
Perinatal Anxiety Screening Scale (PASS) | up to 9 months
  The 31-item PASS is a validated tool for anxiety screening in pregnancy and postpartum.
5-item Primary Care PTSD screen for DSM-5 (PC-PTSD-5) | up to 9 months
  The PC-PTSD-5 is a brief screening tool to identify posttraumatic stress disorder symptom severity.
American Academy of Family Physicians (AAFP) Social Needs Screening Tool | up to 9 months
  Social needs will be assessed with the 14-item American Academy of Family Physicians (AAFP) Social Needs Screening Tool, which includes a range of social determinants of health (housing, food, transportation, utilities, childcare, employment, education, finances, and personal safety).
Recovery Assessment Scale (RAS) | up to 9 months
  Recovery will be measured with the 24-item RAS, a validated tool studied extensively in populations with serious mental illness, which assesses five factors of recovery (personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, and no domination by symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Nichole I Goodsmith, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No